CLINICAL TRIAL: NCT00576342
Title: A Single Dose Patient Preference Study Comparison in Patients With Open-Angle Glaucoma or Ocular Hypertension
Brief Title: Patient Preference Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: C-07-47
Record Dates: First submitted 2007-12-17; First posted 2007-12-19 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — dorzolamide-timolol combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- AL-3862+timolol, then COSOPT (Other): AL-3862+timolol ophthalmic suspension, 1 drop in both eyes, followed by dorzolamide+timolol ophthalmic solution,1 drop in both eyes, 1 day later.
  Interventions: Drug: AL-3862+timolol ophthalmic suspension; Drug: Dorzolamide+timolol ophthalmic solution
- COSOPT, then AL-3862+timolol (Other): Dorzolamide+timolol ophthalmic solution, 1 drop in both eyes, followed by AL-3862+timolol ophthalmic suspension, 1 drop in both eyes, 1 day later.
  Interventions: Drug: AL-3862+timolol ophthalmic suspension; Drug: Dorzolamide+timolol ophthalmic solution

INTERVENTIONS:
Drug: AL-3862+timolol ophthalmic suspension
Drug: Dorzolamide+timolol ophthalmic solution
  Other Names: COSOPT

SUMMARY:
In this randomized crossover study, patients will receive a single drop of two test articles and assess comfort.

ELIGIBILITY:
Inclusion Criteria:

* Sign informed consent;
* Diagnosis of glaucoma or ocular hypertension;
* On a stable regimen of any intraocular pressure (IOP) lowering medication (mono-therapy);
* IOP for which, in the opinion of the investigator, participation in the study does not present a risk to ocular health;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Best corrected visual acuity worse than 0.60 logMAR (20/80 Snellen) in either eye;
* Pregnant, nursing, or not using highly effective birth control methods;
* Use of oral or topical corticosteroids within 30 days of the Screening Visit and during the course of the study;
* History of bronchial asthma or severe chronic obstructive pulmonary disease;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2007-12; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with a stated preference for either study medication | Day 2

SECONDARY OUTCOMES:
Mean ocular discomfort score | Day 1, 1 minute after drop instillation